CLINICAL TRIAL: NCT02547610
Title: MR/PET in the Evaluation of Patients With Esophageal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201402050MINC
Record Dates: First submitted 2015-09-10; First posted 2015-09-11 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Esophageal Cancer
Keywords: MR/PET in the evaluation; patients
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: The imaging biomarkers determined by MR-PET — Combining PET and MRI, namely MR/PET, has the benefit of evaluating tissue metabolism with PET and at the same time evaluating tissue morphology/functional information with MR.

SUMMARY:
In this prospective study, we will recruit newly diagnosed esophageal cancer patients and perform MR/PET before and after chemoradiation therapy. In MR, new image sequences will be added to the conventional sequences, such as high resolution image, DWI, DCE, cine imaging.

DETAILED DESCRIPTION:
Total 80 patients will be recruited and followed after treatment complete for at least two years. We will compare the staging accuracy of MR/PET and PET/CT, and also analyze parameters that are predictive of disease recurrence and patient survival.

ELIGIBILITY:
Inclusion Criteria:

1. newly diagnosed esophageal cancer patient
2. age older than 20 years

Exclusion Criteria:

1. For the safety reason, patients with the following conditions are contraindicated to enter magnetic resonance imaging (MRI) machine due to the high magnetic field, including: cardiac pacemaker, metallic artificial valve, intracranial and mediastinal vascular clips, cardiac defibrillator, nerve stimulator, implanted drug deliver system, metallic foreign body in the eye globe, cochlear implant, metallic fragments in the dangerous body part, Swan-Ganz catheter, and other metallic implants within 8 weeks: such as cardiac valve, stent, coil, filter, and clips.
2. patient who will receive endoscopic local therapy alone
3. unable to finish the standard surgical or radiation treatment
4. history of surgery or radiotherapy to the mediastinum
5. renal insufficiency, contraindication to MR imaging and contrast injection patient who have the severe allergic reaction the Gadollium contrast agent
6. patient who have the claustrophobic symptoms are also not suitable for this MR examination
7. pregnancy or lactating women

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this prospective study, we will recruit newly diagnosed esophageal cancer patients and perform MR/PET before and after chemoradiation therapy.Total 80 patients will be recruited and followed after treatment complete for at least two years.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
The imaging biomarkers determined by MR-PET | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Ting-Fang Shih, M.D., Principal Investigator — Department of Medical Imaging, National Taiwan University Hospital.
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan